CLINICAL TRIAL: NCT03372044
Title: A Phase 1, Open Label Study In Healthy Subjects To Investigate The Pharmacokinetics Of Pf 06865571 Following Single Oral Administration Of Immediate And Modified Release Tablets Compared To Immediate Release Oral Suspension Under Fed Conditions
Brief Title: A Study To Evaluate Different Formulations Of PF-06865571 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C2541003; 2017-003797-14 (EudraCT Number)
Record Dates: First submitted 2017-12-06; First posted 2017-12-13 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: Relative bioavailability; Modified release; Pharmacokinetics
MeSH Terms: interventions — ervogastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PF-06865571 (Experimental): Treatment
  Interventions: Drug: PF-06865571 Immediate release suspension; Drug: PF-06865571 Slow release MR tablets; Drug: PF-06865571 Fast release MR tablets; Drug: PF-06865571 Immediate release tablets

INTERVENTIONS:
Drug: PF-06865571 Immediate release suspension — Suspension
Drug: PF-06865571 Slow release MR tablets — Modified release tablets
Drug: PF-06865571 Fast release MR tablets — Modified release tablets
Drug: PF-06865571 Immediate release tablets — Immediate release tablets

SUMMARY:
An open-label study to understand the effect of different modified release and immediate release formulations on plasma PF-06865571 concentrations after single oral administration under fed conditions

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and female of non-childbearing potential
* Age of 18-55, inclusive
* Body Mass Index 17.5 to 30.5 kg/m2, inclusive
* Body weight >50 kg
* Not on any prescription or non-prescription drugs within 7 days or 5 half-lives prior to first dose.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug test.
* History of regular alcohol consumption exceeding 14 drinks/week for female subjects or 21 drinks/week for male subjects (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).
* Screening supine BP >=140 mm Hg (systolic) or >= 90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Screening supine 12 lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec.
* Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level >=1.25 × upper limit of normal (ULN);
  * Total bilirubin level >=1.5 × ULN; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is =<ULN.
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin induced thrombocytopenia only if heparin is used to flush any intravenous catheters in the study.
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).
* Unwilling or unable to comply with Lifestyle Requirements in the protocol
* Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Subjects who have previously participated in prior studies with PF 06865571 as the investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) for PF-06865571 | 0,0.5,1,2,3,4,6,8,12,24,36,48 hours post dose in each period
Time to Reach Maximum Observed Concentration for PF-06865571 | 0,0.5,1,2,3,4,6,8,12,24,36,48 hours post dose in each period
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06865571 | 0,0.5,1,2,3,4,6,8,12,24,36,48 hours post dose in each period
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time for PF-06865571 | 0,0.5,1,2,3,4,6,8,12,24,36,48 hours post dose in each period
  AUC (0-infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-infinity). It is obtained from AUC (0-t) plus AUC (t-infinity).
Plasma Decay Half-Life (t1/2) for PF-06865571 | 0,0.5,1,2,3,4,6,8,12,24,36,48 hours post dose in each period
  Plasma Decay Half-Life (t1/2)

SECONDARY OUTCOMES:
Number of subjects with adverse events (AEs) | Baseline up to 35 days after last dose
  Number of participants with reported adverse events
Number of subjects with laboratory tests findings of potential clinical importance | Baseline (Day 0) up to 48 hours after last dose of study medication
  Number of participants with potentially clinically important laboratory test findings
Number of subjects with electrocardiogram (ECG) findings of potential clinical importance | Baseline (Day 0) up to 48 hours after last dose of study medication
  Number of participants with potentially clinically important ECG findings
Number of subjects with vital signs findings of potential clinical importance | Baseline (Day 0) up to 48 hours after last dose of study medication
  Number of participants with potentially clinically important vital sign measurements

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C2541003&StudyName=A+Phase+1%2C+Open+Label+Study+In+Healthy+Subjects+To+Investigate+The+Pharmacokinetics+Of+Pf+06865571+Following+Single+Oral+Administration+Of+Immediate+And+Modified+Release+Tablets+Compared+To+Immediate+Release+Oral+Suspension+Under+Fed+Conditions